CLINICAL TRIAL: NCT05348837
Title: Naturalistic Sleep Assessed by Wearable Devices in Parkinson Disease
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0393
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subthalamic nucleus (STN) DBS: Patients undergoing evaluation for subthalamic nucleus DBS implantation will be included in this group.
  Interventions: Procedure: Deep brain stimulation
- Globus pallidus interna (GPi) DBS: Patients undergoing evaluation for globus pallidus interna DBS implantation will be included in this group.
  Interventions: Procedure: Deep brain stimulation

INTERVENTIONS:
Procedure: Deep brain stimulation — Candidacy for DBS implantation will be determined by the treating team, which includes a neurologist, neurosurgeon, neuropsychologist, neuro-radiologist, and palliative care physician.

SUMMARY:
The cardinal motor features of Parkinson's disease (PD) include bradykinesia, rest tremor, and rigidity. Though non-motor features have been recognized for centuries, only recently has the prevalence and impact of non-motor symptoms become the focus of intense study. Disturbances of sleep are among the most common non-motor manifestations of PD; approximately two-thirds of PD patients experience sleep dysfunction of some kind. Given that sleep contributes to the regulation of many physiological processes, sleep disturbance has a significant impact on quality of life in PD, and places high strain on caregivers. Though numerous symptomatic therapies exist, the treatment of sleep disorders in PD is limited by a lack of adequately powered, randomized studies providing high quality evidence. Although deep brain stimulation (DBS) is primarily used to treat PD motor symptoms and reduce the need for dopaminergic medications, several studies have shown that DBS provides benefit for non-motor symptoms, including sleep disturbance. Few studies have used an objective measure to assess the impact of DBS on sleep in PD, and none have done so by studying sleep in the home environment. Existing studies have largely been limited to a single night of sleep recording in a sleep lab. Furthermore, no studies have assessed sleep both on and off medication, before and after DBS implantation. This study will enroll patients undergoing evaluation for DBS implantation. Sleep will be assessed before DBS implantation, both while patients continue their usual medication regimen and while withholding medications. After DBS implantation and programming, sleep will again be assessed with stimulation on, both while continuing medications and subsequently while withholding medications.

ELIGIBILITY:
Inclusion Criteria:

Research subjects must be willing and able to do the following:

* Be able to learn to use and maintain a wristband-style sleep monitor
* Wear a wristband-style sleep monitor for two weeks
* Be able to learn to use and maintain a headband sleep monitor
* Wear a headband sleep monitor for two weeks
* Log daily routine events, such sleeping, eating, and medication regimens for the two-week study period
* Withhold dopaminergic medications after 5:00pm for three consecutive nights

Exclusion Criteria:

Subjects will be excluded if they:

* Carry a diagnosis of dementia (e.g., Parkinson's Disease Dementia or Dementia with Lewy Bodies)
* Currently use or recently (within past 30 days) used a sedative-hypnotic agent for sleep (e.g., Zolpidem, Suvorexant, Eszopiclone)
* Fulfill criteria or carry a diagnosis of a circadian sleep-wake rhythm disorder, as defined by the International Classification of Sleep Disorders, Third Edition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing evaluation for DBS candidacy are eligible to participate in this study. Those deemed appropriate for DBS implantation and who undergo bilateral DBS will complete the second (post-operative) phase of the study. Candidacy for DBS implantation will be determined by the treating team, which includes a neurologist, neurosurgeon, neuropsychologist, neuro-radiologist, and palliative care physician. Decision to participate in the study will have no bearing on DBS candidacy. Patients are eligible to participate in this study regardless of device being implanted.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in total sleep time (TST) as measured by polysomnogram-capable headband | Baseline; 6 months
  The total amount of time spent asleep, averaged over the 3-night study period, will be measured by a polysomnogram-capable headband (Dreem Headband, Rythm, France).

SECONDARY OUTCOMES:
Change in sleep efficiency (SE) as measured by polysomnogram-capable headband | Baseline; 6 months
  SE, defined as the amount of time spent asleep divided by the amount of time spent in bed, averaged over the 3-night study period, will be measured by a polysomnogram-capable headband (Dreem Headband, Rythm, France).
Change in sleep onset latency (SOL) as measured by polysomnogram-capable headband | Baseline; 6 months
  SOL, defined as the amount of time between lying in bed to attempt to sleep and the onset of sleep, averaged over the 3-night study period, will be measured by a polysomnogram-capable headband (Dreem Headband, Rythm, France).
Change in wake after sleep onset (WASO) as measured by polysomnogram-capable headband | Baseline; 6 months
  WASO, defined as the amount of time spent awake after the initial onset of sleep, averaged over the 3-night study period, will be measured by a polysomnogram-capable headband (Dreem Headband, Rythm, France).
Change in total sleep time (TST) as measured by actigraphy | Baseline; 6 months
  Total amount of time spent asleep, averaged over the 3-night study period, will be measured by actigraphy
Change in sleep efficiency (SE) as measured by actigraphy | Baseline; 6 months
  SE, defined as the amount of time spent asleep divided by the amount of time spent in bed, averaged over the 3-night study period, will be measured by actigraphy.
Change in sleep onset latency (SOL) as measured by actigraphy | Baseline; 6 months
  SOL, defined as the amount of time between lying in bed to attempt to sleep and the onset of sleep, averaged over the 3-night study period, will be measured by actigraphy.
Change in wake after sleep onset (WASO) as measured by actigraphy | Baseline; 6 months
  WASO, defined as the amount of time spent awake after the initial onset of sleep, averaged over the 3-night study period, will be measured by actigraphy.

OTHER OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) score | Baseline; 6 months
  The PSQI is a well-validated clinical questionnaire that queries subjects on seven sleep parameters.
Change in Parkinson Disease Sleep Scale, version 2 (PDSS-2) score | Baseline; 6 months
  The PDSS-2 is a 15-item scale which specifically queries several sleep disturbances commonly afflicting PD patients, including restless leg syndrome, nocturia, pain, and sleep apnea
Change in Fatigue Severity Scale (FSS) score | Baseline; 6 months
  The FSS is a nine-item scale that measures the severity of fatigue and its impact on daily life.
Change in Epworth Sleepiness Scale (ESS) score | Baseline; 6 months
  The ESS is a self-administered, eight-item assessment of daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Baumgartner, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR